CLINICAL TRIAL: NCT05322993
Title: Improving Polyp Detection Rate by Artificial Intelligence in Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haraldsplass Deaconess Hospital (Other)
Collaborators: Haukeland University Hospital (Other); European Society of Gastrointestinal Endoscopy (Other); Kanalspesialistene AS (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: REK 275068
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Colonic Polyp
Keywords: Colonoscopy; Artificial intelligence; Polyp detection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Endoscopists will perform colonoscopies in three consecutive phases; 1. without artificial intelligence (AI), 2. with AI, 3. without (AI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With artificial intelligence (AI) (Active Comparator): Use of GI Genius artificial intelligence device during colonoscopy.
  Interventions: Device: GI Genius
- Without artificial intelligence (Active Comparator): Use of standard colonoscopy equipment without GI Genius.
  Interventions: Device: Standard white light colonoscope

INTERVENTIONS:
Device: GI Genius — The use of artificial intelligence during colonoscopy to improve polyp detection.
  Arms: With artificial intelligence (AI)
Device: Standard white light colonoscope — Standard colonoscopy.
  Arms: Without artificial intelligence

SUMMARY:
The aim of this study is to investigate if the use of artificial intelligence (AI) in colonoscopy improves the polyp detection rate, and if the use of AI has a learning effect.

DETAILED DESCRIPTION:
The endoscopists will use GI Genius from Medtronic, a device that uses artificial intelligence (AI) based on machine learning to detect polyps in the colon in real time during colonoscopy. The device interprets the endoscopy pictures and superimposes possible polyps with frames.

The patients will be included in regular outpatient clinics in Western Norway. The endoscopists will be divided into groups depending on their experience. The endoscopists will perform colonoscopies in three phases; (1) before the use of AI, (2) during the use of AI and (3) after the use of AI. The investigators will then evaluate the polyp detection rate (PDR) in the three phases to see if AI increases PDR, and if there is a learning effect on PDR after the use of AI. The investigators will also evaluate if there is a difference in the learning-effect from AI-use depending on if the endoscopist is experienced or inexperienced.

The PDR's are registered as part of Norway's national quality register of colonoscopy, Gastronet. The data registered in Gastronet can also help the investigators evaluate other outcomes such as withdrawal time, bowel preparation, patient reported pain, patient satisfaction and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming to outpatient clinics to perform colonoscopies

Exclusion Criteria:

* Total colectomy
* Reservation against registration in Gastronet, the national quality register for colonoscopy in Norway

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5034 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Polyp detection rate (PDR) with and without artificial intelligence (AI) | 18 months
  Evaluate the PDR with and without the use of GI Genus artificial intelligence
PDR after the use of AI, is there a learning effect? | 18 months
  Evaluate if there is an improved PDR after the use of AI

SECONDARY OUTCOMES:
Withdrawal time | 18 months
  To evaluate if the withdrawal time is influenced by the use of artificial intelligence
Complications | 24 months
  To evaluate if there are more registered complications with the use of AI

CONTACTS AND LOCATIONS:
Overall Officials: Roald F. Havre, Professor, Study Director — Helse Bergen
Locations (3):
- Norway (3):
  - Haraldsplass Deaconess Hospital, Bergen, Vestland
  - Haukeland University Hospital, Bergen, Vestland
  - Kanalspesialistene AS, Bergen, Vestland

IPD SHARING:
Plan to Share IPD: No
There is no specific plan to share IPD with other researchers.

REFERENCES:
- See also: Gastronet, the national quality register of colonoscopies — https://www.sthf.no/gastronet